CLINICAL TRIAL: NCT07370207
Title: A Phase 2 Multi-center, Randomized, Open-label Study to Assess the Efficacy and Safety of AHB-137 in Nucleos(t)Ide Analogue-treated Participants With HBeAg Negative Chronic Hepatitis B in the Asia Pacific Region
Brief Title: Phase 2 Study of AHB-137 in HBeAg Negative Chronic Hepatitis B (CHB) Participants in Asia Pacific Region
Acronym: ASPIRE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AusperBio Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB-10-8011
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis; Chronic Hepatitis; Chronic Hepatitis B; Hepatitis B; Hepatitis B, Chronic; Hepatitis B Virus; hepatitis B virus e-antigen; AHB-137; Nucleos(t)ide analog; Nucleos(t)ide analogue; Antisense Oligonucleotide; Blood-Borne Infections; Communicable Diseases; Infections; DNA Virus Infections; Virus Diseases; Hepatitis, Viral, Human; Liver Diseases; Digestive System Diseases; Chronic Disease; Disease Attributes; Pathologic Processes; Pathological Conditions, Signs and Symptoms
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis; Hepatitis, Chronic; Hepatitis B; Blood-Borne Infections; Communicable Diseases; Infections; DNA Virus Infections; Virus Diseases; Hepatitis, Viral, Human; Liver Diseases; Digestive System Diseases; Chronic Disease; Disease Attributes; Pathologic Processes; Pathological Conditions, Signs and Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: AHB-137 + 2 LDs (Experimental): AHB-137 300 mg subcutaneous (SC) weekly for 24 weeks with 2 loading doses (LDs) on Days 4 and 11
  Interventions: Drug: AHB-137
- Arm B: AHB-137 + 3 LDs (Experimental): AHB-137 300 mg SC weekly for 24 weeks with 3 LDs on Days 4, 11, and 18
  Interventions: Drug: AHB-137

INTERVENTIONS:
Drug: AHB-137 — Subcutaneous injection

SUMMARY:
This study is a randomized, open-label, multicenter phase 2 clinical trial to evaluate the efficacy and safety of AHB-137 injection in participants with HBeAg-negative CHB treated with NAs.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Adults ≥18 years of age (or per local age of majority) and ≤65 years of age at Screening who are able to provide informed consent, comply with study procedures, and agree to discontinue nucleos(t)ide analog (NA) therapy if protocol-defined discontinuation criteria are met.
2. Body mass index (BMI) ≤35 kg/m².
3. Documented chronic hepatitis B virus (HBV) infection for ≥6 months prior to randomization, defined by hepatitis B surface antigen (HBsAg) positivity or detectable HBV DNA.
4. Hepatitis B e antigen (HBeAg) negative at Screening.
5. Receiving stable, approved nucleos(t)ide analog (NA) monotherapy for ≥6 months prior to randomization.
6. HBV DNA below the lower limit of quantification (LLOQ) at Screening.
7. Hepatitis B surface antigen (HBsAg) level >100 IU/mL and ≤3,000 IU/mL at Screening.
8. Alanine aminotransferase (ALT) ≤2 × upper limit of normal (ULN) at Screening.
9. Screening electrocardiogram (ECG) without clinically significant abnormalities and with a Fridericia-corrected QT interval (QTcF) ≤450 msec for males or ≤470 msec for females.
10. Females of childbearing potential must not be breastfeeding and must have a negative serum pregnancy test at Screening and a negative urine pregnancy test prior to first dose.
11. Male and female participants of childbearing potential must agree to use protocol-specified effective contraception during the dosing period and for ≥6 months after the last dose of AHB-137.

Exclusion Criteria:

Participants will be excluded from the study if any of the following criteria apply:

1. Clinically significant disease other than chronic hepatitis B virus (HBV) infection, as documented in medical history or identified on physical examination, including but not limited to acute coronary syndrome within 6 months prior to Screening, significant or unstable cardiac disease, uncontrolled diabetes, bleeding diathesis or coagulopathy, or prior solid organ or bone marrow transplant
2. Concomitant clinically significant liver disease, including but not limited to viral hepatitis caused by other pathogens, hemochromatosis, Wilson's disease, primary biliary cholangitis, autoimmune liver disease, alcoholic liver disease, drug-induced liver injury, or current or prior history of clinical hepatic decompensation (e.g., ascites, encephalopathy, hepatorenal syndrome, or variceal hemorrhage).
3. Any severe infection (other than chronic HBV infection) within 1 month prior to randomization and/or requiring intravenous anti-infective therapy.
4. History of immune thrombocytopenia.
5. Current suspected liver cirrhosis and/or evidence of cirrhosis defined as liver stiffness measurement (LSM) >9 kPa by FibroScan® or equivalent imaging modality (e.g., ultrasound elastography).
6. History of liver cirrhosis defined by liver biopsy or by LSM >12 kPa by FibroScan® or equivalent imaging modality.
7. Prior history of, current diagnosis of, or suspected hepatocellular carcinoma (HCC), or alpha-fetoprotein (AFP) ≥20 ng/mL at Screening.
8. History of extrahepatic diseases potentially associated with HBV infection, including but not limited to nephrotic syndrome, any form of glomerulonephritis, polyarteritis nodosa, cryoglobulinemia, or uncontrolled hypertension.
9. Laboratory evidence of active infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis D virus (HDV), or active syphilis. Participants with positive HCV or HDV serology and documented negative HCV RNA or HDV RNA, respectively, are eligible.
10. Abnormal laboratory values at Screening meeting any of the following criteria:

    1. Serum albumin <3.5 g/dL
    2. Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m² calculated using the CKD-EPI equation (or JSN-CKDI equation for participants in Japan)
    3. International normalized ratio (INR) >1.25
    4. Platelet count <125 × 10⁹/L
    5. Total bilirubin >1.5 × upper limit of normal (ULN). Participants with benign unconjugated hyperbilirubinemia (Gilbert's syndrome) may be enrolled if deemed eligible by the Investigator
    6. Urine albumin-to-creatinine ratio (uACR) >0.3 mg/mg (300 mg/g) on two consecutive measurements following a positive or weakly positive urine protein result on routine urinalysis
    7. Borderline positive or positive antineutrophil cytoplasmic antibody (ANCA) results requiring further evaluation (MPO-ANCA and PR3-ANCA). Eligibility requires review of complete medical history and confirmation of no past or current vasculitic, inflammatory, or autoimmune disease by the Sponsor or Sponsor-designated Medical Monitor
11. History of vasculitis or presence of signs or symptoms suggestive of vasculitis (e.g., vasculitic rash, skin ulceration, unexplained recurrent hematuria), or history or presence of diseases associated with vasculitis (e.g., systemic lupus erythematosus, rheumatoid arthritis, relapsing polychondritis, mononeuritis multiplex).
12. History of malignancy within 5 years prior to Screening, except for adequately treated non-melanoma skin cancer. Participants currently undergoing evaluation for potential malignancy are excluded.
13. History of hypersensitivity or allergy to any component of the investigational product (IP).
14. Major trauma or major surgery within 3 months prior to Screening, or planned surgery during the study period unless eligibility is confirmed by the Medical Monitor.
15. Current alcohol or substance abuse that, in the Investigator's judgment, may interfere with study participation or compliance.
16. Female participants who are pregnant, breastfeeding, planning pregnancy during the study, or unwilling to refrain from egg donation and/or in vitro fertilization during the study.
17. Participation in another clinical trial or receipt of any investigational product prior to first dose in this study within:

    1. Five half-lives (if known) or twice the duration of biological effect (if known), whichever is longer, or
    2. Six months, if neither half-life nor duration of effect is known
18. Prior treatment with antisense oligonucleotides (ASOs) or small interfering RNA (siRNA)-based therapies.
19. Any of the following prior or concomitant therapies:

    1. Prolonged use of immunomodulators (e.g., corticosteroids, methotrexate), cytotoxic drugs, or biologics (e.g., monoclonal antibodies) within 6 months prior to first IP administration, except for short-term treatment (≤2 weeks) or topical/inhaled corticosteroids
    2. Interferon therapy within 12 months prior to first dose
    3. Vaccination within 1 month prior to Screening, except for influenza or SARS-CoV-2 (COVID-19) vaccination or booster
    4. Current treatment with bulevirtide
20. Requirement for long-term regular use of anticoagulants (e.g., warfarin, factor Xa inhibitors) or antiplatelet agents (e.g., clopidogrel or regular aspirin), except for low-dose aspirin, unless the Investigator determines the medication can be safely discontinued prior to first IP administration. Participants taking low-dose aspirin must agree to discontinue use during the study if protocol-specified conditions are met.
21. Any other condition or circumstance that, in the Investigator's judgment, would make the participant unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with sustained response post AHB-137 treatment | 24 Weeks post AHB-137 treatment
  Sustained response defined as hepatitis B surface antigen (HBsAg) level below the limit of detection (LOD, 0.05 international units [IU]/mL) and HBV deoxyribonucleic acid (DNA) below the lower limit of quantification (LLOQ)

SECONDARY OUTCOMES:
Proportion of participants with functional cure (FC) or sustained HBV DNA response off all HBV treatment | Off-treatment follow-up (Week 48 to 96)
Proportion of participants with functional cure (FC) | Week 72
Proportion of participants with sustained HBV DNA response | From baseline through Week 72
Proportion of participants with HBsAg ≤10 IU/mL and HBV DNA < Lower Limit of Quantification (LLOQ) post AHB-137 treatment | 24 weeks post AHB-137 treatment
Proportion of participants with HBsAg <100 IU/mL and HBV DNA < LLOQ | 24 weeks post AHB-137 treatment and at Week 72
Proportion of participants with complete response (CR) | From baseline through end of study (Week 96)
Proportion of participants with HBsAg < or ≥ LOD (0.05 IU/mL) and/or HBV DNA < or ≥ LLOQ | From baseline through end of study (Week 96)
Proportion of participants with ultrasensitive HBsAg < LOD (0.005 IU/mL) | From baseline through end of study (Week 96)
Proportion of participants with HBsAg ≤ 10 IU/mL and < 100 IU/mL | From baseline through end of study (Week 96)
Proportion of participants that meet nucleos(t)ide analog (NA) discontinuation criteria | Week 48
Categorical change from baseline in serum hepatitis B surface antigen (HBsAg) levels, defined as reductions of ≥0.5, ≥1.0, ≥1.5, ≥2.0, or ≥3.0 log₁₀ IU/mL, assessed at each scheduled study visit | From baseline through end of study (Week 96), assessed at each scheduled visit
Proportion of participants with anti-HBs seroconversion (with hepatitis B surface antibody [HBsAb] > 10 IU/L) | Weeks 24, 48, and 72
Quantitative hepatitis B virologic and serologic markers over time | From baseline through end of study (Week 96)
  Actual values and change from baseline over time in quantitative hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAb), hepatitis B virus (HBV) DNA, HBV ribonucleic acid (RNA), hepatitis B core-related antigen (HBcrAg), hepatitis B e antibody (HBeAb), and hepatitis B e antigen (HBeAg), summarized descriptively.
Proportion of participants who experience virologic relapse | From baseline through Week 72
Time from nucleos(t)ide analog (NA) therapy discontinuation to virologic relapse | From NA therapy discontinuation (Week 48) through end of follow-up (Week 96)
Change from baseline in alanine aminotransferase (ALT) | From baseline through end of study (Week 96)
Proportion of participants with baseline ALT above the upper limit of normal (ULN) who achieve ALT normalization | From baseline through end of study (Week 96)
Proportion of patients with drug-resistant mutations | From baseline through end of study (Week 96)
Proportion of participants with treatment-emergent adverse events (TEAEs) | From first dose (Day 1) through end of study (Week 96)
  Proportion of participants who experience treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and adverse events leading to discontinuation of study treatment.
Proportion of participants with detectable anti-drug antibody (ADA) to AHB-137 and corresponding ADA titers | From baseline through end of study (Week 96)
Area under the plasma concentration-time curve (AUC) of AHB-137 | From first dose (Day 1) through end of pharmacokinetic sampling (Week 48)
Concentration at the end of the dosing interval (Ct) of AHB-137 | From first dose (Day 1) through end of pharmacokinetic sampling (Week 48)
Maximum observed plasma concentration (Cmax) of AHB-137 | From first dose (Day 1) through end of pharmacokinetic sampling (Week 48)
Time to maximum observed plasma concentration (Tmax) of AHB-137 | From first dose (Day 1) through end of pharmacokinetic sampling (Week 48)
Apparent plasma clearance (CL/F) of AHB-137 | From first dose (Day 1) through end of pharmacokinetic sampling (Week 48)
Population Pharmacokinetic and Exposure-Response Analyses of AHB-137 | From first dose (Day 1) through end of study (Week 96)
  Population pharmacokinetic modeling of AHB-137, including covariate analysis and assessment of exposure-response relationships for pharmacodynamic, efficacy, and safety endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Lau, MD, PhD, Study Chair — AusperBio Therapeutics Inc.
Locations (8):
- St Vincents Hospital Melbourne, Fitzroy, Victoria, Australia
- Queen Mary Hospital - PPDS, Hong Kong, China
- New Zealand Clinical Research, Grafton, Auckland, New Zealand
- National University Hospital - Singapore, Singapore, Singapore
- Asan Medical Center, Seoul, South Korea
- Taiwan (3):
  - Chiayi Christian Hospital, Chiayi City
  - E-DA Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No